CLINICAL TRIAL: NCT05227118
Title: A Randomized Clinical Study to Evaluate the Safety and Tolerability of MK-8189 in Participants With Alzheimer's Disease With or Without Symptoms of Agitation-Aggression and/or Psychosis
Brief Title: MK-8189 Safety and Tolerability in Participants With Alzheimer's Disease With or Without Symptoms of Agitation-Aggression and/or Psychosis (MK-8189-017)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8189-017; MK-8189-017 (Other: Merck)
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — MK-8189

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-8189 (Experimental): Participants will be assigned to one of the following regimens: Titration 1: 4 mg x 2 tablets Days 1-3; 4 mg x 1 tablet & 12 mg x 1 tablet Days 4-28 OR Titration 2: 4 mg x 2 tablets Days 1-3; 4 mg x 1 tablet & 12 mg x 1 tablet Days 4-6; 12 mg x 2 tablets Days 7-28 OR Titration 3: 4 mg x 1 tablet Days 1-3; 4 mg x 2 tablets Days 4-6; 4 mg x 1 tablet & 12 mg x 1 tablet Days 7-9; 12 mg x 2 tablets Days 10-28.
  Interventions: Drug: MK-8189
- Placebo (Placebo Comparator): Participants will be assigned to one of the following regimens: Titration 1: 2 tablets Days 1-28 OR Titration 2: 2 tablets Days 1-28 OR Titration 3: 1 tablet Days 1-3; 2 tablets Days 4-28.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8189 — MK-8189 administered orally once a day (QD) at a titration via tablet in 4 mg and 12 mg dose strengths
  Arms: MK-8189
Drug: Placebo — MK-8189 matching placebo administered orally QD
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple ascending doses of MK-8189 in participants with Alzheimer's Disease (AD) with or without symptoms of agitation-aggression and/or psychosis.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has a documented diagnosis of probable Alzheimer Disease based on National Institute on Aging-Alzheimer Association criteria for AD, with a history of cognitive and functional decline with gradual onset and slow progression for at least 1 year before screening, that is either corroborated by an informant who knows the participant well or is documented in medical records
* Lives in the community setting with a reliable trial partner/caregiver or lives alone in an assisted living facility, with supervision and has a reliable trial partner/caregiver
* Has a reliable and competent trial partner/caregiver who must have a close relationship with the participant and is knowledgeable of the participant's condition and progress and able to read, understand and speak the designated language at the study site
* Can read at the 6th grade level/equivalent as determined by the investigator
* Has an academic and/or employment history sufficient to exclude intellectual disability and is able, in the opinion of the investigator, to fully participate in the study
* Participants receiving treatment with a cholinesterase inhibitor or other treatment for AD, must have been on a stable regimen for 3 months prior to screening and there are no expected changes in co-medication during the study
* Is able to discontinue any antipsychotic medication they are taking at the time of Screening
* Has a body mass index (BMI) > 18 and ≤ 35kg/m2, inclusive

Exclusion Criteria:

* Has agitation/aggression or psychosis that is attributable to concomitant medications, environmental conditions, substance abuse, or an active medical or psychiatric condition
* Has a known history of stroke or evidence from prior magnetic resonance imaging (MRI) scan (if available) that is clinically important in the investigator's opinion
* Has evidence of a clinically relevant neurological disorder other than the disease being studied (i.e., probable AD) at Screening
* Has a history of seizures or epilepsy within the last 5 years before Screening
* Has evidence of a clinically relevant or unstable psychiatric disorder
* Is at imminent risk of self-harm
* Has a history of alcoholism or drug dependency/abuse within the last 5 years before Screening
* Has a history of cancer (malignancy). Exceptions: (1) Adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix or; (2) Other malignancies that have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study
* Has a family history of long QT syndrome
* Previously developed severe extrapyramidal symptoms (EPS) following administration of any prescribed medication or study treatment
* Is positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV)
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pre-study (screening) visit
* Consumes greater than 3 glasses of alcoholic beverages per day
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* Is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 3 years

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (8):
- United States (8):
  - CITrials ( Site 0007), Santa Ana, California
  - Top Medical Research ( Site 0005), Cutler Bay, Florida
  - Velocity Clinical Research, Hallandale Beach ( Site 0001), Hallandale, Florida
  - Well Pharma Medical Research, Corp. ( Site 0006), Miami, Florida
  - Atlanta Center for Medical Research ( Site 0004), Atlanta, Georgia
  - iResearch Atlanta ( Site 0009), Decatur, Georgia
  - Global Medical Institutes LLC; Princeton Medical Institute ( Site 0008), Princeton, New Jersey
  - Richmond Behavioral Associates ( Site 0003), Staten Island, New York

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 8 sites in the United States.
Groups:
- Titration 1: MK-8189: Participants received MK-8189 8 mg on Days 1 to 3 and MK-8189 16 mg on Days 4 to 28 during Titration 1.
- Titration 1: Placebo: Participants received placebo matched to MK-8189 during Titration 1.
- Titration 2: MK-8189: Participants received MK-8189 8 mg on Days 1 to 3, 16 mg on Days 4 to 6, and 24 mg on Days 7 to 28 during Titration 2.
- Titration 2: Placebo: Participants received placebo matched to MK-8189 during Titration 2.
Period: Overall Study
Arm/Group | Titration 1: MK-8189 | Titration 1: Placebo | Titration 2: MK-8189 | Titration 2: Placebo
Started | 6 | 2 | 16 | 5
Completed | 6 | 2 | 13 | 5
Not Completed | 0 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Titration 1: MK-8189 | Titration 1: Placebo | Titration 2: MK-8189 | Titration 2: Placebo | Total
Number analyzed (Participants) | 6 | 2 | 16 | 5 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (4.0) | 71.5 (0.7) | 71.6 (7.6) | 71.2 (4.5) | 71.7 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 7 | 3 | 15
  Male | 3 | 0 | 9 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 11 | 5 | 22
  Not Hispanic or Latino | 2 | 0 | 5 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 5 | 0 | 9
  White | 4 | 0 | 11 | 5 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Results are reported according to dose.
Time Frame: Up to approximately 42 days
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Groups:
- MK-8189 8 mg: Participants received MK-8189 8 mg on Days 1 to 3 during Titrations 1 and 2.
- MK-8189 16 mg: Participants received MK-8189 16 mg on Days 4 to 28 during Titration 1, and on Days 4 to 6 during Titration 2.
- MK-8189 24 mg: Participants received MK-8189 24 mg on Days 7 to 28 during Titration 2.
- Placebo: Participants received placebo matched to MK-8189 during Titrations 1 and 2.
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Placebo
Number analyzed (Participants) | 22 | 22 | 14 | 7
Participants | 3 | 8 | 5 | 1

2. Primary Outcome: Number of Participants Discontinuing From Study Therapy Due to AE
Description: as for outcome 1
Time Frame: Up to approximately 42 days
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Placebo
Number analyzed (Participants) | 22 | 22 | 14 | 7
Participants | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 42 days
Description: All participants are included.
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/14 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/22 | 0/14 | 0/7
Other Adverse Events (participants affected / at risk) | 3/22 | 8/22 | 5/14 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8189 8 mg (N=22) | MK-8189 16 mg (N=22) | MK-8189 24 mg (N=14) | Placebo (N=7)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK-8189 8 mg (N=22) | MK-8189 16 mg (N=22) | MK-8189 24 mg (N=14) | Placebo (N=7)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Electric shock sensation (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT05227118/Prot_SAP_000.pdf